CLINICAL TRIAL: NCT02665195
Title: Prospective Registry of Multiplex Testing (PROMPT): Phase II
Brief Title: Prospective Registry of Multiplex Testing (PROMPT)
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Mayo Clinic (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 16-017
Record Dates: First submitted 2016-01-20; First posted 2016-01-27 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Genetic Testing
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Biospecimen Retention: Samples With DNA — saliva specimen

GROUPS / COHORTS (1):
- Prospective Registry of Multiplex Testing: This is a prospective ascertainment study that will obtain medical information and biospecimens from two different types of families: 1) Families transmitting sequence variants in non-BRCA predisposition genes that are either functionally deleterious or likely to be functionally deleterious based upon the interpretation of the laboratory that performed the testing on the Index Participant (Initial PROMPT enrollee), and 2) Families transmitting variants of uncertain significance (usually rare missense variants) in non- BRCA predisposition genes. Attempts will be made to collect a biospecimen and a completed risk factor questionnaire from each participant.
  Interventions: Other: saliva specimen; Behavioral: questionnaire

INTERVENTIONS:
Other: saliva specimen
Behavioral: questionnaire

SUMMARY:
This study is being done to learn more about how changes in certain genes may be linked to cancer. Some people with cancer got their disease because they inherited an abnormal (mutated) gene.

The researchers of this study want to better understand the risks that are linked to genetic changes in these less well-studied genes. By understanding these risks, we believe that doctors will be able to give better advice to families with mutations in these genes.

DETAILED DESCRIPTION:
PROMPT (Prospective Registry of Multiplex Testing) is an Internet-based, patient-directed ascertainment study. It is a partnership between Memorial Sloan Kettering, University of Pennsylvania, Mayo Clinic, and Dana Farber Cancer Institute in collaboration with Ambry Genetics, GeneDx, Myriad Genetics, Pathway Genomics, and Quest Laboratories (5 laboratories providing multiplex panel testing commercially).

ELIGIBILITY:
Inclusion Criteria:

* Individual with deleterious (pathogenic) or likely deleterious (likely pathogenic) mutation in a cancer susceptibility gene OR
* Individual with a variant of uncertain significance (VUS) in a cancer susceptibility gene OR
* Family members, either tested or not tested, who are part of a family known to be transmitting a deleterious or likely deleterious mutation or a variant of uncertain significance in a cancer predisposition gene

Exclusion Criteria:

* Inability or refusal to participate in consent discussion
* Subject is less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be conducted as a multi-center study with the involvement of attendings, genetic counselors, and research study staff at the participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 689 (Actual)
Dates: Start 2016-01; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Acquire DNA samples | 3 years
Acquire pathology materials | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Robson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering @ Rockville, Rockville Centre, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/